CLINICAL TRIAL: NCT03834532
Title: Living Well After Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Ohio State University (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Michael P Pignone, Professor of Medicine, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-05-0009
Record Dates: First submitted 2019-01-28; First posted 2019-02-08 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer Female; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer; Ductal Carcinoma in Situ; Ductal Breast Carcinoma; Lobular Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Carcinoma, Lobular

STUDY DESIGN:
Intervention Model Description: Participants enrolled in the study will complete a baseline survey. Participants will then be randomized to receive a breast reconstruction decision aid or an educational website on healthy living with breast cancer. Participants will complete a second survey after viewing the assigned material. Participants may be invited to complete a third survey six months after surgery.
Who Masked: Participant
Masking Description: Participants enrolled in the study will complete a baseline survey. Participants will then be randomized to receive a breast reconstruction decision aid or an educational website on healthy living with breast cancer. Participants will complete a second survey after viewing the assigned material. Participants may be invited to complete a third survey six months after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants randomized to the intervention group will receive a breast reconstruction decision aid. Participants will be provided instructions on how to access and navigate the decision aid. Participants will access the decision aid through a website link that is emailed to them or on a tablet at the study site.
  Interventions: Other: Breast reconstruction decision aid
- Control (Active Comparator): Participants randomized to the control group will receive two website pages on healthy living with breast cancer from an educational website. Participants will be provided instructions on how to access and navigate the website pages. Participants will access the website pages through a link that is emailed to them or on a tablet at the study site.
  Interventions: Other: Educational website

INTERVENTIONS:
Other: Breast reconstruction decision aid — The breast reconstruction decision aid is a web-based, interactive tool that participants will use after the first breast surgery visit and before a plastic surgery visit or surgery. The decision aid provides information about post-mastectomy breast reconstruction and helps the participant clarify their preferences related to the procedure.
  Other Names: Web-based tool
  Arms: Intervention
Other: Educational website — The educational website contains information on healthy living with breast cancer including, physical activity and nutrition.
  Other Names: Website
  Arms: Control

SUMMARY:
Decision making about whether to have breast reconstruction after mastectomy can be difficult, and previous studies have found that many women are not well informed about their options. Patient decision aids can improve decision quality for a variety of health conditions. This pilot randomized study seeks to determine how a patient decision aid about breast reconstruction affects the quality of decisions about reconstruction including patient knowledge, concordance between preferences and treatment, and decisional regret.

DETAILED DESCRIPTION:
Enrolled participants will be randomized to 1 of 2 arms; participants may receive a breast reconstruction decision aid or an educational website on healthy living with breast cancer.

Participants will complete up to three surveys; a baseline survey before viewing the decision aid or website, a second survey immediately after viewing the decision aid or website, and a third survey six months after surgery. Tablets will be made available to participants at the study site through which they can complete the surveys and view the decision aid or website. Participants will have the options of viewing the decision aid or website outside of the study site, and completing the three surveys electronically or on paper.

The baseline survey and second survey will each take approximately 45 minutes for participants to complete. The third survey will take approximately 30 minutes for participants to complete.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Adult (18 years or older)
* New diagnosis of incident or recurrent Stage I-III ductal or lobular carcinoma, or Ductal Carcinoma in Situ (DCIS)
* Not yet had mastectomy
* Considering or planning to have mastectomy
* Able to read and speak English
* Competent to make health care decisions

Exclusion Criteria:

* Male
* Age less than 18 years
* Diagnosis of stage IV breast cancer, inflammatory breast cancer, phyllodes, or sarcoma
* Already had mastectomy for this diagnosis
* Planning to have breast conservation therapy
* Not being treated by a Texas Oncology surgeon or oncologist
* Not able to read and speak English
* Not competent to make health care decisions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Number of patients enrolled per month | 12 months
  To determine the feasibility of recruiting eligible patients and delivering the breast reconstruction decision support intervention. Measured by the number of patients enrolled per month.
Proportion of patients retained at 6 months | 6 months
  To determine the feasibility of recruiting eligible patients and delivering the breast reconstruction decision support intervention. Measured by the proportion of patients retained through the 6 month outcome assessment.

SECONDARY OUTCOMES:
How a patient decision aid about breast reconstruction affects knowledge about reconstruction. | 6 months
  Change in knowledge (e.g. advantages and disadvantages) about breast reconstruction from baseline to post intervention measured by Decision Quality Instrument - Reconstruction Module.
How a patient decision aid about breast reconstruction affects concordance of patient values and decisions about reconstruction. | 6 months
  Concordance between preferences (e.g. concerns about appearance, complications, recovery) regarding breast reconstruction and treatment outcome (mastectomy with immediate breast reconstruction, mastectomy without immediate breast reconstruction) at 6-month follow-up measured by Rating Scale.
How a patient decision aid about breast reconstruction affects concordance of patient values and decisions about reconstruction. | 6 months
  Concordance between preferences (e.g. concerns about appearance, complications, recovery) regarding breast reconstruction and treatment outcome (mastectomy with immediate breast reconstruction, mastectomy without immediate breast reconstruction) at 6-month follow-up measured by Ranking Task.
How a patient decision aid about breast reconstruction affects concordance of patient values and decisions about reconstruction. | 6 months
  Concordance between preferences (e.g. concerns about appearance, complications, recovery) regarding breast reconstruction and treatment outcome (mastectomy with immediate breast reconstruction, mastectomy without immediate breast reconstruction) at 6-month follow-up measured by Decisional Conflict Scale.
How a patient decision aid about breast reconstruction affects concordance of patient values and decisions about reconstruction. | 6 months
  Concordance between preferences (e.g. concerns about appearance, complications, recovery) regarding breast reconstruction and treatment outcome (mastectomy with immediate breast reconstruction, mastectomy without immediate breast reconstruction) at 6-month follow-up measured by treatment outcome recorded in patient electronic health record (EHR).
How a patient decision aid about breast reconstruction affects decision making outcomes. | 6 months
  Regret with decision related to breast reconstruction at 6-month follow-up measured by Decisional Regret Scale.
How a patient decision aid about breast reconstruction affects decision making outcomes. | 6 months
  Satisfaction with decision related to breast reconstruction at 6-month follow-up measured by Satisfaction with Decisions Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Oncology, Austin, Texas, United States